CLINICAL TRIAL: NCT03512379
Title: Clinical Trial for the Application of Robotic System in Spinal Surgery: a Randomized Controlled Study
Brief Title: Clinical Trial for the Application of Robotic System in Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Wei Tian, Professor, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JST-201508
Record Dates: First submitted 2018-04-03; First posted 2018-04-30 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Robotic Surgical Procedures; Spinal Surgery; Safety
Keywords: robot-assisted surgery; pedicle screw; spine
MeSH Terms: interventions — Fluoroscopy

STUDY DESIGN:
Intervention Model Description: Robot-assisted surgery group Free-hand surgery group Navigation-assisted surgery group
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Robot assisted surgery group (Experimental): Spinal surgery using TIANJI Robot system.
  Interventions: Device: TIANJI Robot
- Free hand surgery group (Active Comparator): Spinal surgery using fluoroscopy-based free hand technique
  Interventions: Device: Fluoroscopy
- Navigation-assisted surgery group (Active Comparator): Spinal surgery using Navigation-assisted technique
  Interventions: Device: Navigation

INTERVENTIONS:
Device: TIANJI Robot — A robotic system for spinal surgery
  Arms: Robot assisted surgery group
Device: Fluoroscopy — For fluoroscopy-based free hand surgery
  Arms: Free hand surgery group
Device: Navigation — For navigation-assisted spinal surgery
  Arms: Navigation-assisted surgery group

SUMMARY:
This randomized controlled study was designed to evaluate the accuracy, safety and clinical outcomes of the robot assisted spinal surgery.

DETAILED DESCRIPTION:
Robot assisted operation is new for spinal surgery, in this study, we will evaluate the accuracy, safety and clinical outcomes compared with traditional free hand operation and navigation assisted operation.

ELIGIBILITY:
Inclusion Criteria:

* Spinal disease required for screw fixation；signed the inform consent

Exclusion Criteria:

* Patients with severe osteoporosis; patients with old fractures; patients with pedicle deformity; patients with severe systemic diseases; patients with coagulation disorders; patients who are considered unsuitable for this trail by the clinician.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Screw guide wire adjustment times | During surgery
  The adjustment times of screw guide wire during surgery
Screw adjustment times | During surgery
  The adjustment times of screw during surgery
Deviation of screw | Up to 12 weeks
  The deviation between the actual position of screw and the preoperative designed position
Perforation rate of screw | Up to 12 weeks
  Rate of screws breaching out pedicles on postoperative CT image

SECONDARY OUTCOMES:
Operation time | During surgery
  Operation time
Blood loss | During surgery
  Blood loss during surgery
Complications | Up to 4 weeks
  Complications after surgery
Hospital stay after surgery | Up to 4 weeks
  Hospital stay after surgery
Hospitalization costs | Up to 4 weeks
  Hospitalization costs
Visual Analogue Scale | 3 days before surgery
  Visual Analogue Scale
Visual Analogue Scale | 3 days after surgery
  Visual Analogue Scale
Neck Disability Index | 3 days before surgery
  Neck Disability Index
Neck Disability Index | 3 days after surgery
  Neck Disability Index
Oswestry Disability Index | 3 days before surgery
  Oswestry Disability Index
Oswestry Disability Index | 3 days after surgery
  Oswestry Disability Index
modified Japanese orthopaedic association score | 3 days before surgery
  modified Japanese orthopaedic association score
modified Japanese orthopaedic association score | 3 days after surgery
  modified Japanese orthopaedic association score

CONTACTS AND LOCATIONS:
Overall Officials: Wei Tian, MD,PHD, Study Chair — Beijing Jishuitan Hospital
Locations (1):
- Beijing Jishuitan Hospital, Beijing, Beijing Municipality, China